CLINICAL TRIAL: NCT01841112
Title: Safety, Tolerability and Pharmacokinetics of Single Oral Doses of BI 409306 (Tablet) in Healthy Chinese and Japanese Male Volunteers and Multiple Oral Doses of BI 409306 (Tablet) in Healthy Japanese Male Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 409306 Tablets in Healthy Asian Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.4
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Results first posted 2024-05-28 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Healthy

ARMS (5):
- Placebo (Placebo Comparator): Subjects received matching placebo to the BI-409306 (film-coated tablet/s), administered orally on day 1 for single dose (SD) segment and on day 3 to day 9 for multiple dose (MD) segment
  Interventions: Drug: Placebo
- BI-409306 25 milligram (mg) SD (Experimental): Subjects received 25 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
  Interventions: Drug: BI-409306 25 milligram (mg) SD
- BI-409306 50 mg SD (Experimental): Subjects received 50 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
  Interventions: Drug: BI-409306 50 mg SD
- BI-409306 100 mg SD (Experimental): Subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
  Interventions: Drug: BI-409306 100 mg SD
- BI-409306 100 mg MDBI-409306 100 mg SD & MD (Experimental): Subjects received 100 mg multiple dose of BI-409306 (film-coated tablet/s), administered orally once on day 3 to day 9. A wash-out period of 48 hours was included before the second dose (first does of multipled dose segment) was administered. Subjects were considered for both single dose (following first dose) and multiple dose purposes.
  Interventions: Drug: BI-409306 100 mg MD

INTERVENTIONS:
Drug: Placebo — Subjects received matching placebo to the BI-409306 (film-coated tablet/s), administered orally on day 1 for single dose (SD) segment and on day 3 to day 9 for multiple dose (MD) segment
  Arms: Placebo
Drug: BI-409306 25 milligram (mg) SD — Subjects received 25 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
  Arms: BI-409306 25 milligram (mg) SD
Drug: BI-409306 50 mg SD — Subjects received 50 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
  Arms: BI-409306 50 mg SD
Drug: BI-409306 100 mg SD — Subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
  Arms: BI-409306 100 mg SD
Drug: BI-409306 100 mg MD — Subjects received 100 mg multiple dose of BI-409306 (film-coated tablet/s), administered orally once on day 3 to day 9
  Arms: BI-409306 100 mg MDBI-409306 100 mg SD & MD

SUMMARY:
Safety, tolerability and pharmacokinetics of single and multiple oral doses of BI 409306 tablets in healthy Chinese and Japanese male volunteers of a known genotype as specified in the study protocol.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male Chinese and Japanese volunteers
2. Age between 20 and 45 years
3. BMI between 18.5 and 25 kg/m2 (Body Mass Index)
4. Known genotype as specified in the study protocol
5. Subjects must be able to understand and comply with study requirements

Exclusion criteria:

1. Any deviation from healthy condition

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2013-07-18 (Actual); Study Completion 2013-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.4.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was randomised, placebo controlled and double-blind within dose groups, single dose (3 dose groups), multiple dose (1 dose group, 8-day treatment), single centre trial with healthy Chinese and Japanese male volunteers
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI-409306 100 mg SD & MD: Subjects received 100 mg multiple dose of BI-409306 (film-coated tablet/s), administered orally once on day 3 to day 9. A wash-out period of 48 hours was included before the second dose (first dose of multiple dose segment) was administered. Subjects were considered for both single dose (following first dose) and multiple dose purposes.
Period: Single Dose Segment (Day 1)
Arm/Group | Placebo | BI-409306 25 Milligram (mg) SD | BI-409306 50 mg SD | BI-409306 100 mg SD | BI-409306 100 mg SD & MD
Started | 16 | 12 | 12 | 19 | 6
Completed | 15 | 11 | 11 | 19 | 6
Not Completed | 1 | 1 | 1 | 0 | 0
Not completed — Not Treated | 1 | 1 | 1 | 0 | 0
Period: Washout (48 Hours)
Arm/Group | Placebo | BI-409306 25 Milligram (mg) SD | BI-409306 50 mg SD | BI-409306 100 mg SD | BI-409306 100 mg SD & MD
Started | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Multiple Dose Segment (Days3-9)
Arm/Group | Placebo | BI-409306 25 Milligram (mg) SD | BI-409306 50 mg SD | BI-409306 100 mg SD | BI-409306 100 mg SD & MD
Started | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) included all randomised subjects who were documented to have received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI-409306 25 Milligram (mg) SD | BI-409306 50 mg SD | BI-409306 100 mg SD | BI-409306 100 mg SD & MD | Total
Number analyzed (Participants) | 15 | 11 | 11 | 19 | 6 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.9 (3.1) | 26.5 (4.0) | 26.6 (6.4) | 27.4 (5.8) | 26.3 (2.9) | 26.4 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 11 | 11 | 19 | 6 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 11 | 11 | 19 | 6 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Poor metaboliser (PM) / extensive metaboliser (EM) [Count of Participants; unit: Participants] — Number of subjects per category: Poor metaboliser (PM) / extensive metaboliser (EM).
  Participants
    Poor metaboliser (PM) | 4 | 0 | 0 | 6 | 6 | 16
    Extensive metaboliser (EM) | 11 | 11 | 11 | 13 | 0 | 46
Ethnicity [Count of Participants; unit: Participants]
  Chinese | 8 | 5 | 6 | 13 | 0 | 32
  Japanese | 7 | 6 | 5 | 6 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Subjects With Drug-related Adverse Events (AEs)
Description: Percentage (%) of subjects with drug-related adverse events (AEs).
Time Frame: From first drug administration until 11 days after last dose of study medication, up to 18 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Groups:
- BI-409306 100 mg MD-PM: Subjects received 100 mg multiple dose of BI-409306 (film-coated tablet/s), administered orally once on day 3 to day 9 in multiple dose (MD) segment
- BI-409306 100 mg SD-PM: Subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1 in multiple dose (MD) segment
Arm/Group | Placebo | BI-409306 25 Milligram (mg) SD | BI-409306 50 mg SD | BI-409306 100 mg SD | BI-409306 100 mg MD-PM | BI-409306 100 mg SD-PM
Number analyzed (Participants) | 15 | 11 | 11 | 19 | 6 | 6
Percentage of Participants | 13.3 | 9.1 | 36.4 | 57.9 | 83.3 | 83.3

2. Secondary Outcome: Maximum Measured Concentration of a Single Dose of BI 409306 in Plasma (Cmax)
Description: Maximum measured concentration of a single dose of BI 409306 in plasma (Cmax).
Time Frame: PK plasma samples: 2 hours before drug administration and 10, 20, 30, 45 minutes, 1, 1:30, 2, 2:30, 3, 4, 6, 8, 10, 12, 14, 24 hours for SD segment after drug administration.
Population: The pharmacokinetic set (PKS) included all subjects of the treated set who provided at least one evaluable observation for at least one pharmacokinetic (PK) endpoint without Important protocol violation (IPV) that could potentially influence the results of PK measurements for determination of primary PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) / Litre (L)
Groups:
- BI-409306 25 mg - Chinese: 5 Chinese EM subjects received 25 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 50 mg - Chinese: 6 Chinese EM subjects received 50 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 100 mg - Chinese: 7 Chinese EM subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 100 mg - Chinese (PM): 6 Chinese PM subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 25 mg - Japanese: 6 Japanese EM subjects received 25 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 50 mg - Japanese: 5 Japanese EM subjects received 50 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 100 mg - Japanese: 6 Japanese EM subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
- BI-409306 100 mg SD & MD - Japanese (PM): Subjects received 100 mg multiple dose of BI-409306 (film-coated tablet/s), administered orally once on day 3 to day 9. A wash-out period of 48 hours was included before the second dose (first dose of multiple dose segment) was administered. Subjects were considered for both single dose (following first dose) and multiple dose purposes.
  For the current endpoint only data collected following the first dose were considered.
Arm/Group | BI-409306 25 mg - Chinese | BI-409306 50 mg - Chinese | BI-409306 100 mg - Chinese | BI-409306 100 mg - Chinese (PM) | BI-409306 25 mg - Japanese | BI-409306 50 mg - Japanese | BI-409306 100 mg - Japanese | BI-409306 100 mg SD & MD - Japanese (PM)
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 6 | 5 | 6 | 6
nanomol (nmol) / Litre (L) | 292 (113.0) | 824 (74.1) | 1970 (77.8) | 4020 (26.8) | 496 (26.5) | 914 (32.5) | 3290 (43.0) | 4510 (26.8)
Statistical Analysis 1: Comparison: BI-409306 25 mg - Chinese vs BI-409306 50 mg - Chinese vs BI-409306 100 mg - Chinese vs BI-409306 100 mg - Chinese (PM); Dose proportionality was assessed in Chinese subjects. For the power model perfect dose proportionality would correspond to a slope of 1; Test type: Superiority or Other; Slope = 1.3712, 95% CI 2-sided [0.7272 to 2.0151] — The standard error of slope estimate = 0.3038
Statistical Analysis 2: Comparison: BI-409306 25 mg - Japanese vs BI-409306 50 mg - Japanese vs BI-409306 100 mg - Japanese vs BI-409306 100 mg SD & MD - Japanese (PM); Dose proportionality was assessed in Japanese subjects. For the power model perfect dose proportionality would correspond to a slope of 1; Test type: Superiority or Other; Slope = 1.3652, 95% CI 2-sided [1.0421 to 1.6883] — The standard error of slope estimate = 0.1516

3. Secondary Outcome: Area Under the Concentration-time Curve of a Single Dose of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of a single dose of BI 409306 in plasma over the time interval from 0 extrapolated to infinity (AUC 0-infinity).
Time Frame: as for outcome 2
Population: The pharmacokinetic set (PKS) included all subjects of the treated set who provided at least one evaluable observation for at least one pharmacokinetic (PK) endpoint without Important protocol violation (IPV) that could potentially influence the results of PK measurements for determination of primary PK endpoints. Only subjects with non missing values were included in the endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Arm/Group | BI-409306 25 mg - Chinese | BI-409306 50 mg - Chinese | BI-409306 100 mg - Chinese | BI-409306 100 mg - Chinese (PM) | BI-409306 25 mg - Japanese | BI-409306 50 mg - Japanese | BI-409306 100 mg - Japanese | BI-409306 100 mg SD & MD - Japanese (PM)
Number analyzed (Participants) | 5 | 5 | 7 | 6 | 6 | 5 | 6 | 6
nanomol (nmol) * hour (h) / Litre (L) | 376 (67.7) | 1070 (119.0) | 2020 (106.0) | 7550 (21.4) | 504 (24.7) | 985 (40.3) | 2100 (47.1) | 8650 (32.1)
Statistical Analysis 1: Comparison: BI-409306 25 mg - Chinese vs BI-409306 50 mg - Chinese vs BI-409306 100 mg - Chinese vs BI-409306 100 mg - Chinese (PM); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Slope = 1.1998, 95% CI 2-sided [0.4794 to 1.9202] — The standard error of slope estimate = 0.3380
Statistical Analysis 2: Comparison: BI-409306 25 mg - Japanese vs BI-409306 50 mg - Japanese vs BI-409306 100 mg - Japanese vs BI-409306 100 mg SD & MD - Japanese (PM); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Slope = 1.0299, 95% CI 2-sided [0.7131 to 1.3466] — The standard error of slope estimate = 0.1486

4. Secondary Outcome: Area Under the Concentration-time Curve of a Single Dose of BI 409306 in Plasma Over the Time Interval 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of a single dose of BI 409306 in plasma over the time interval 0 to the last quantifiable data point (AUC0-tz).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Arm/Group | BI-409306 25 mg - Chinese | BI-409306 50 mg - Chinese | BI-409306 100 mg - Chinese | BI-409306 100 mg - Chinese (PM) | BI-409306 25 mg - Japanese | BI-409306 50 mg - Japanese | BI-409306 100 mg - Japanese | BI-409306 100 mg SD & MD - Japanese (PM)
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 6 | 5 | 6 | 6
nanomol (nmol) * hour (h) / Litre (L) | 375 (67.8) | 1040 (102.0) | 2020 (106.0) | 7550 (21.4) | 504 (24.8) | 985 (40.3) | 2100 (47.1) | 8640 (32.1)
Statistical Analysis 1: Comparison: BI-409306 25 mg - Chinese vs BI-409306 50 mg - Chinese vs BI-409306 100 mg - Chinese vs BI-409306 100 mg - Chinese (PM); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Slope = 1.2015, 95% CI 2-sided [0.5078 to 1.8952] — The standard error of slope estimate = 0.3272
Statistical Analysis 2: Comparison: BI-409306 25 mg - Japanese vs BI-409306 50 mg - Japanese vs BI-409306 100 mg - Japanese vs BI-409306 100 mg SD & MD - Japanese (PM); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Slope = 1.0301, 95% CI 2-sided [0.7133 to 1.3469] — The standard error of slope estimate = 0.1486

5. Secondary Outcome: Maximum Measured Concentration of the Metabolite CD 13896 in Plasma (Cmax)
Description: Maximum measured concentration of the metabolite CD 13896 in plasma (Cmax) after single administration of BI 409306.
Time Frame: as for outcome 2
Population: The pharmacokinetic set (PKS) included all subjects of the treated set who provided at least one evaluable observation for at least one pharmacokinetic (PK) endpoint without Important protocol violation (IPV) that could potentially influence the results of PK measurements for determination of primary PK endpoints. As pre-specified in the protocol, metabolite analyses were only planned for the 100 mg extensive metabolizer groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) / Litre (L)
Groups:
- BI-409306 100 mg - Chinese: 6 Chinese EM subjects received 100 mg single dose of BI-409306 (film-coated tablet/s), administered orally once on day 1
Arm/Group | BI-409306 100 mg - Chinese | BI-409306 100 mg - Japanese
Number analyzed (Participants) | 6 | 6
nanomol (nmol) / Litre (L) | 926 (30.9) | 1080 (24.5)

6. Secondary Outcome: Maximum Measured Concentration of the Metabolite CD 14084 in Plasma (Cmax)
Description: Maximum measured concentration of the metabolite CD 14084 in plasma (Cmax) after single administration of BI 409306.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) / Litre (L)
Arm/Group | BI-409306 100 mg - Chinese | BI-409306 100 mg - Japanese
Number analyzed (Participants) | 6 | 6
nanomol (nmol) / Litre (L) | 3800 (21.8) | 4340 (16.9)

7. Secondary Outcome: Area Under the Concentration-time Curve of the Metabolite CD 13896 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of the metabolite CD 13896 in plasma over the time interval from 0 extrapolated to infinity (AUC 0-infinity) after single administration of BI 409306.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Arm/Group | BI-409306 100 mg - Chinese | BI-409306 100 mg - Japanese
Number analyzed (Participants) | 6 | 6
nanomol (nmol) * hour (h) / Litre (L) | 1650 (14.2) | 1520 (15.6)

8. Secondary Outcome: Area Under the Concentration-time Curve of the Metabolite CD 14084 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of the metabolite CD 14084 in plasma over the time interval from 0 extrapolated to infinity (AUC 0-infinity) after single administration of BI 409306.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Arm/Group | BI-409306 100 mg - Chinese | BI-409306 100 mg - Japanese
Number analyzed (Participants) | 6 | 6
nanomol (nmol) * hour (h) / Litre (L) | 8670 (10.8) | 9060 (14.6)

9. Secondary Outcome: Area Under the Concentration-time Curve of the Metabolite CD 13896 in Plasma Over the Time Interval 0 to the Last Quantifiable Data Point (AUC0-tz).
Description: Area under the concentration-time curve of the metabolite CD 13896 in plasma over the time interval 0 to the last quantifiable data point (AUC0-tz) after single administration of BI 409306.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Arm/Group | BI-409306 100 mg - Chinese | BI-409306 100 mg - Japanese
Number analyzed (Participants) | 6 | 6
nanomol (nmol) * hour (h) / Litre (L) | 1650 (14.2) | 1510 (15.6)

10. Secondary Outcome: Area Under the Concentration-time Curve of the Metabolite CD 14084 in Plasma Over the Time Interval 0 to the Last Quantifiable Data Point (AUC0-tz).
Description: Area under the concentration-time curve of the metabolite CD 14084 in plasma over the time interval 0 to the last quantifiable data point (AUC0-tz) after single administration of BI 409306.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Arm/Group | BI-409306 100 mg - Chinese | BI-409306 100 mg - Japanese
Number analyzed (Participants) | 6 | 6
nanomol (nmol) * hour (h) / Litre (L) | 8670 (10.8) | 9060 (14.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until 11 days after last dose of study medication, up to 18 days.
Description: Treated Set (TS) included all randomised subjects who were documented to have received at least one dose of study medication.
Arm/Group | Placebo | BI-409306 25 Milligram (mg) SD | BI-409306 50 mg SD | BI-409306 100 mg SD | BI-409306 100 mg SD-PM | BI-409306 100 mg MD-PM
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11 | 0/11 | 0/19 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/15 | 1/11 | 5/11 | 11/19 | 5/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | BI-409306 25 Milligram (mg) SD (N=11) | BI-409306 50 mg SD (N=11) | BI-409306 100 mg SD (N=19) | BI-409306 100 mg SD-PM (N=6) | BI-409306 100 mg MD-PM (N=6)
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 4 | 1 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 3 | 1 | 1
Photopsia (Eye disorders) | 0 | 0 | 1 | 5 | 2 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.